CLINICAL TRIAL: NCT03403348
Title: A Randomized, Double-blind, Placebo-controlled, First-in-human, 6-Part Study of Orally Administered JNJ-64417184 to Evaluate the Safety, Tolerability, and Pharmacokinetics of Single and Multiple Ascending Doses, and the Antiviral Activity of Multiple Doses in a Respiratory Syncytial Virus (RSV) Challenge Study in Healthy Subjects
Brief Title: A First-In-Human Study of Orally Administered JNJ-64417184 to Evaluate the Safety, Tolerability, and Pharmacokinetics of Single and Multiple Ascending Doses, and the Antiviral Activity of Multiple Doses in a Respiratory Syncytial Virus (RSV) Challenge Study in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen BioPharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: JNJ-184-1401; 2017-004363-13 (EudraCT Number); JNJ-184-1401 (Other: Janssen Biopharma, Inc.)
Record Dates: First submitted 2017-12-21; First posted 2018-01-18 (Actual); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Part 1: Single Ascending Dose (SAD) (Experimental): Participants will be enrolled in 7 cohorts and receive one of the 7 corresponding SADs of JNJ-64417184, starting from 40 milligram (mg), or placebo in a fasted state. Dose escalation in the subsequent cohorts will depend on the human maximum observed plasma concentration (Cmax) and area under the plasma concentration-time curve (AUC) in previous cohorts.
  Interventions: Drug: JNJ-64417184; Drug: Placebo
- Part 2A: Food Effect (Experimental): Participants enrolled in cohort 4 of part 1 will roll-over in Part 2A and will receive a single oral dose (the same dose as received in Part 1) of JNJ-64417184 or placebo with a high-fat meal.
  Interventions: Drug: JNJ-64417184; Drug: Placebo
- Part 2B: Relative Bioavailability (Optional) (Experimental): Participants enrolled in cohorts 5, 6, 7 or any other optional cohorts of Part 1 will roll-over in Part 2B and will receive a single oral dose (the same dose as received in Part 1) of JNJ-64417184 or placebo under fasted state. Dosing may be changed from fasted to a fed state, depending on emerging pharmacokinetics (PK) data from Part 2A.
  Interventions: Drug: JNJ-64417184; Drug: Placebo
- Part 3: Multiple Ascending Dose (MAD) (Experimental): Participants will be enrolled in 3 cohorts and will receive one of the 3 corresponding MADs of JNJ-64417184 or placebo, dosed once daily for 7 days. There will be 3 optional cohorts and participants in these cohorts will follow 7- to 14-day dosing schedule. Dosing will either occur in the fasted or the fed state, depending on the outcome of Part 2A. Dose selection and dose escalation in the MAD cohorts will depend on the observed human Cmax and AUC in previous (SAD) cohorts. Additional cohorts may be evaluated at the discretion of the Sponsor and the Principal Investigator (PI).
  Interventions: Drug: JNJ-64417184; Drug: Placebo
- Part 4: Human RSV Challenge (Proof-of-Concept Study Part) (Experimental): Based on emerging PK and safety data from Part 3 (MAD), the participants inoculated with respiratory syncytial virus (RSV) -A Memphis 37b and confirmed positive by polymerase chain reaction (PCR) will either receive JNJ-64417184 or placebo once daily OR receive JNJ-64417184 (low dose), JNJ-64417184 (high dose) or placebo once daily.
  Interventions: Drug: JNJ-64417184; Drug: Placebo
- Part 5: SAD/Japanese (Experimental): Participants of Japanese descent will be enrolled in 3 cohorts and will receive one of the corresponding SADs of JNJ-64417184 or placebo in a fasted state. Dosing may be changed from fasted to a fed state, depending on emerging PK data from Part 2A. The starting dose and formulation will be selected based on the outcome of Parts 1 and 2. Dose escalation in the subsequent cohorts will depend on the observed human Cmax and AUC in previous cohorts.
  Interventions: Drug: JNJ-64417184; Drug: Placebo
- Part 6: MAD/Japanese (Optional) (Experimental): Participants of Japanese descent may be enrolled in 3 cohorts and will receive one of the corresponding MADs of JNJ-64417184 or placebo, dosed once daily for 7 to 14 days. Dosing will either occur in the fasted or the fed state, depending on the outcome of Part 2A. Dose selection and dose escalation in the MAD cohorts will depend on the observed human Cmax and AUC in previous (Parts 1, 2, 3, and 5) cohorts.
  Interventions: Drug: JNJ-64417184; Drug: Placebo

INTERVENTIONS:
Drug: JNJ-64417184 — Participants will receive JNJ-64417184 in Parts 1, 2A, 2B, 3, 4, 5 and 6.
Drug: Placebo — Participants will receive matching placebo to JNJ-64417184 in Parts 1, 2A, 2B, 3, 4, 5 and 6.

SUMMARY:
The purpose of the study is to evaluate the safety and tolerability of single and multiple oral doses of JNJ-64417184 administered to healthy participants and the antiviral effect of multiple oral doses of JNJ-64417184 compared to placebo in participants infected through inoculation with respiratory syncytial virus (RSV)-A Memphis 37b (Part 4).

ELIGIBILITY:
Inclusion Criteria:

* Participant has provided written consent
* In the Investigator's opinion, the participant is able to understand and comply with protocol requirements, instructions, and protocol-stated restrictions and is likely to complete the study as planned
* Participant is in good health as deemed by the Investigator, based on the findings of a medical evaluation including medical history, physical examination, laboratory tests, and electrocardiogram (ECG). In case of an out-of-range clinical laboratory test, vital sign, or ECG value that will determine a participant's eligibility, a retest can be done. Results of this retest must be available prior to the first administration of the study drugs (Parts 1, 3, 5, and 6) or prior to inoculation (Part 4). The result of the retest will be considered for participant eligibility
* Body mass index (BMI) of 18 to 30 kilogram per meter square (kg/m^2) (inclusive), minimum weight of 50 kilogram (kg)
* A female participant is eligible to participate in this study if she is of non childbearing potential defined as either (i) premenopausal with a documented tubal ligation, bilateral oophorectomy, or hysterectomy; or (ii) postmenopausal defined by 12 months of spontaneous amenorrhea and follicle-stimulating hormone level within the laboratory's reference range for postmenopausal females. A postmenopausal female who is receiving hormone replacement therapy and who is willing to discontinue hormone therapy from 28 days before study drug dosing (Parts 1, 3, 5, and 6) or before inoculation (Part 4), and for the entire duration of the study, may be eligible for study participation. A male participant is eligible to participate in this study if (i) he is either surgically sterile or, (ii) in case of having a female partner of childbearing potential, the male participant and partner are practicing and willing to continue to practice highly effective forms of birth control until 90 days after the end of the study. Irrespective of the partner's form of birth control, a male participant must wear a condom when engaging in any activity that allows for passage of ejaculate to another person

Exclusion Criteria:

* Clinically significant cardiovascular, respiratory, renal, gastrointestinal, hematologic, neurologic, endocrinologic, oncologic, ophthalmologic, musculoskeletal, psychiatric or any other uncontrolled medical illness
* Positive human immunodeficiency virus (HIV), active hepatitis A virus (HAV), hepatitis B virus (HBV), or hepatitis C virus (HCV) test
* Creatinine clearance less than (<) 60 milliliter per minute (mL/min) (Cockcroft-Gault)
* Drug allergy such as, but not limited to, allergy to penicillins, including allergies experienced in previous studies with experimental drugs
* Any condition that, in the opinion of the Investigator, would compromise the study or the well-being of the participant or prevent the participant from meeting the study requirements

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 130 (Actual)
Dates: Start 2018-05-09 (Actual); Primary Completion 2019-11-24 (Actual); Study Completion 2019-11-24 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events (AEs) as a Measure of Safety and Tolerability | Approximately up to 8 months
  An AE is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship.
Number of Participants With Laboratory Abnormalities | Approximately up to 8 months
  Number of participants with laboratory abnormalities will be reported.
Number of Participants With Clinically Significant Changes in Vital Signs | Approximately up to 8 months
  Number of participants with clinically significant changes in vital signs will be reported.
Number of Participants With Clinically Significant Changes in Physical Examination Findings | Approximately up to 8 months
  Number of participants with clinically significant changes in physical examination findings will be reported.
Number of Participants With ECG Abnormalities | Approximately up to 8 months
  Number of participants with electrocardiogram (ECG) abnormalities will be reported.
Change From Baseline in QT Interval Corrected According to Fridericia's Formula (QTcF) (Parts 1 and 3) | Baseline up to Day 31
  The QT interval corrected for heart rate (QTc interval) using Fridericia method will be measured by electrocardiograms (ECG) triplicates.
Change From Baseline in Forced Expiratory Volume in 1 Second (FEV1) Absolute as Measured by Spirometry (Part 4) | Baseline up to Day 31
  FEV1 is the amount of air that can be exhaled in one second. FEV1 will be measured by spirometry. A positive change from baseline in absolute FEV1 indicates improvement in lung function.
Change From Baseline in Forced Vital Capacity (FVC) Absolute as Measured by Spirometry (Part 4) | Baseline up to Day 31
  FVC is a standard pulmonary function test used to quantify respiratory muscle weakness. FVC is the volume of air that can forcibly be blown out after full inspiration in the upright position, in liters and will be measured by spirometry.
Change From Baseline in Percent-Predicted FEV1 (Part 4) | Baseline up to Day 31
  FEV1 is the amount of air, measured in liters, forcibly exhaled in 1 second. Pulmonary function tests will be performed by participants in the morning before dosing. The percent predicted FEV1 equals the participant's observed FEV1 divided by the participant's predicted FEV1 (determined by height and race) and converted to a percentage by multiplying by 100 percent (%).
Change From Baseline in Percent-Predicted FVC (Part 4) | Baseline up to Day 31
  Predicted FVC is based on a formula using sex, age and height of a person, and is an estimate of healthy lung capacity. Percent of predicted FVC = (observed value)/(predicted value) * 100 %.
Area Under the Concentration-Time Curve Between Time of First Administration and Dosing Day 7 (AUC[0-Dosing Day 7]) of RSV-A Memphis 37b Viral Load in Participants Infected Through Inoculation With This Viral Strain (Part 4) | Up to Day 7
  Area under the concentration-time curve between time of first administration and Dosing Day 7 (AUC[0-Dosing Day 7)] of respiratory syncytial virus (RSV)-A Memphis 37b viral load in participants infected through inoculation with this viral strain, as determined by a quantitative real-time polymerase chain reaction (qRT PCR) assay of nasal wash (Part 4) will be assessed.

SECONDARY OUTCOMES:
JNJ-64417184 Plasma Concentrations | Approximately up to 67 days
  Plasma concentration of JNJ-64417184 after a single oral dose and after multiple oral doses will be assessed.
JNJ-64417184 Urine Concentrations | Approximately up to 67 days
  Urine concentration of JNJ-64417184 after a single oral dose and after multiple oral doses will be assessed.
Corrected QT Interval (QTc) Duration (Parts 1 and 3) | Up to Day 2 (Part 1); Up to Day 8 (Part 3)
  QTc duration (as calculated from Holter extracts) after a single oral dose and after multiple oral doses administered to healthy participants will be reported.
AUC(0-Dosing Day 7) of RSV Viral Load From Treatment Onset (Part 4) | Up to Day 7
  The AUC(0-Dosing Day 7) of RSV viral load from treatment onset, as determined by a qRT-PCR assay of nasal wash samples and by cell culture (plaque assay) will be reported.
Time to Non-Detectability of RSV (Part 4) | Up to Day 31
  Time to non-detectability of RSV as determined by a qRT-PCR assay of nasal wash samples and by cell culture (plaque assay) will be reported.
Peak RSV Viral Load by Dosing Day (Part 4) | Up to Day 31
  Peak RSV viral load by dosing day as determined by a qRT-PCR assay of nasal wash samples and by cell culture (plaque assay) will be reported.
AUC(0-Dosing Day 7) of Total RSV Symptoms From Treatment Onset | Up to Day 7
  The AUC(0-Dosing Day 7) of total RSV symptoms from treatment onset, using self reported symptoms on the symptom diary card (SDC) will be reported. Participants will assess any challenge virus-related symptoms using the symptom questionnaire in the SDC which will report the symptoms experienced by the participants at the moment on a scale of 0 to 3 where '0' implies 'no symptom' and '3' implies 'bothersome most or all of the time, stopping from participating in activities' OR 'less severe' to 'more severe' symptoms.
Total Weight of Mucus (Part 4) | Up to Day 12
  The total weight of mucus produced from treatment onset will be reported.
Change From Baseline in the RSV L Protein-Encoding Gene Sequence After Treatment (Part 4) | Baseline up to Day 11
  Change from baseline in sequence of the RSV L protein encoding gene before and after treatment, for participants who show rebound, partial viral suppression or non-response to JNJ-64417184, will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Biopharma, Inc. Clinical Trial, Study Director — Janssen BioPharma, Inc.
Locations (2):
- United Kingdom (2):
  - hVIVO Services Limited, London
  - Hammersmith Medicines Research Ltd, London